# Official Title of the Study:

WIC Infant and Toddler Feeding Practices Study-2 (Feeding My Baby, A National WIC Study)

**NCT Number:** 

NCT02031978

Document Date: June 30, 2014

Uploaded 05/15/2021





# Appendix Y.1 Infant Toddler Feeding Study Core Sample Consent form - ENGLISH

#### **Background**

Westat, along with our partners at University of California Los Angeles, Altarum Institute, and University of California Berkeley, is carrying out The *Feeding My Baby* Study for the Food and Nutrition Service of the U.S. Department of Agriculture. About half the babies born in the U.S. are on WIC, and the study is being done to learn more about the choices WIC families make in feeding their children. We are looking for about 4,500 WIC families to take part in our study. We would like you to help by joining the study, and allowing us to hear more about you, your family, and the choices you make in feeding your baby.

# What Would I Do in the Study?

# Take Part in Telephone Interviews

If you agree to participate in this study we will contact you regularly by phone to interview you. If you are pregnant right now, we'd like to interview you once during your pregnancy. We'll also interview you by phone up to ten times during your baby's first two years. Interviews will take place every other month during the first year starting about when your baby is one month old (or starting at three months if your baby is already more than one month old). During your child's second year we'll interview you when your child is thirteen months, fifteen months, eighteen months, and twenty-four months old. The interviews will ask you about your background, your household, your experiences in WIC, your health and your child's health, the choices you make about how and what to feed your baby, your beliefs and advice you've gotten about feeding babies and toddlers, and your family's and child's behavior and habits. Each interview will take about thirty minutes.

#### Allow Us to Seek WIC Records

We will, with your permission, seek WIC record information about you and your child several times over the course of the study. This will include information on the food packages WIC gives you or your child, and your child's weight and length. If we lose touch with you, we might also ask WIC for information on how to contact you.

#### Allow Us to Seek Birth Hospital Records

We will, with your permission, seek information about your baby's birth from the hospital where you gave birth. This will include your baby's health at birth, any complications at birth, and how your baby was fed in the hospital.

According to the Paperwork Reduction Act of 1995, no persons are required to respond to a collection of information unless it displays a valid OMB number. The valid OMB control number for this information collection is 0584-0580. The time required to complete this information collection is estimated to average 5 minutes per response, including the time for reviewing instructions, searching existing data sources, gathering and maintaining the data needed, and completing and reviewing the collection of information.

If Necessary, Allow Us to Seek a Health Professional's Measures of Child Length and Weight As long as you remain in WIC, we will get information about your child's length and weight from WIC. But if you stop going to WIC we will ask your permission to get length and weight from either your child's doctor, or if your child hasn't seen a doctor, from a study nurse who will make arrangements with you to come measure and weigh your child.

## What Are the Risks of Being In This Study?

We expect that your time in the study will be interesting and pleasant, and will not cause you discomfort. We will take many steps and precautions to protect your privacy. Your name and your child's name will not be used in any research reports. We will assign a study ID to your information, and only a small number of study staff will have access to the connection between study IDs and actual names. All study information will be stored on secure computer servers at Westat. We will not share personal information about you with WIC or with anyone else who is not on the study staff.

# What Are the Benefits of Being In This Study?

There are no direct benefits to you for taking part in this study. The information collected during the study will help the Food and Nutrition Service understand better how WIC mothers choose to feed their babies and toddlers, and how WIC services help mothers with those choices. They will then use this information to continue to improve WIC services for everyone.

To thank you for the time you take to be in this study, we will offer you a prepaid MasterCard with \$50 sent by mail within two weeks after you join for this first introduction to the study, and \$20 for every interview you complete after that.

### What Are My Rights As a Participant In the Study?

Taking part in this study is completely voluntary. Giving consent means that you have heard or read the information about this study and that you agree to take part. You may still decide not to answer any questions we ask that you don't want to answer. If you decide not to take part in an interview, we will continue to get records from WIC about you for the rest of the study period unless you tell us to stop that as well. If you decide to take part in the study and then change your mind, you can stop at any time. There is no penalty for stopping taking part in the study, and it won't affect any WIC services or other benefits you otherwise get.

#### Who Should I Call if I Have Questions?

If you have questions about the study itself and what we are doing, a member of our study team can help you. For those questions, please contact #NAME at XXX-XXXXXXX.

If you have a problem that the study team member couldn't help you resolve, please call Dr. Gail Harrison at 310-825-3738.

| If you have questions about you | our rights as | a participant | in this | study, | please | contact | Sharon | Zack, |
|---|---|---|---|---|---|---|---|---|
| the Westat IRB Administrator | , at 1-800-93 | 37-8281. | | | | | | |

By signing below, I am saying that I have heard or read the information presented here, and I agree to take part in the Feeding My Baby study.

| Signature |
|---|
| Date |
| If the person signing above is not yet a legal adult, please see below: |
| By signing below, I am saying that I have heard or read the information presented here, and as a parent or legal guardian I give permission for the person signing above to take part in the Feeding My Baby study. |
| Signature |
| Date |